CLINICAL TRIAL: NCT05032976
Title: A Prospective, Single-arm, Open-label, Non-interventional, Multicenter to Assess the Safety of BNT162b2 in Domestic Post-marketing Surveillance
Brief Title: Korea Comirnaty Post-marketing Surveillance
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4591025; NCT05032976 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: COVID-19; Vaccines; Adverse Effects; SARS-CoV-2; Safety
Keywords: COVID-19; Vaccines,; Adverse Effects; SARS-CoV-2; Safety
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine; Aging; famtozinameran

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Tozinameran (BNT162b2): Subjects aged 6 months and older who are scheduled for Tozinameran vaccination
  Interventions: Biological: Tozinameran 12 Years of age and older; Biological: Tozinameran 5 to 11 Years of age; Biological: Tozinameran 6 months to 4 years of age
- Riltozinameran (BNT162b2 OMI BA.1): Subject aged 12 years and older who are scheduled for Riltozinameran vaccination
  Interventions: Biological: Riltozinameran 12 Years of age and older
- Famtozinameran (BNT162b2 OMI BA.4-5): Subject aged 5 years and older who are scheduled for Famtozinameran vaccination
  Interventions: Biological: Famtozinameran 12 Years of age and older; Biological: Famtozinameran 5 to 11 Years of age
- Raxtozinameran (BNT162b2 OMI XBB.1.5): Subject aged 6 months to 4 years and 12 years and older who are scheduled for Raxtozinameran vaccination
  Interventions: Biological: Raxtozinameran 12 years of age and older; Biological: Raxtozinameran 6 months to 4 years of age

INTERVENTIONS:
Biological: Tozinameran 12 Years of age and older — BNT162b2 (purple cap) is administered with dilution, while BNT162b2 (grey cap) is administered without dilution. Both formulations are administered by intramuscular injection (IM) of 0.3 mL. According to the approved and authorized label, the recommended dose of BNT162b2 is a series of two doses (1 day 1 dose, 0.3mL each) 21 days apart and administered IM.
  Groups: Tozinameran (BNT162b2)
Biological: Tozinameran 5 to 11 Years of age — BNT162b2 (orange cap) is administered with dilution by intramuscular injection (IM) of 0.2mL. According to the approved and authorized label, the recommended dose of BNT126b2 is a series of two dose (1day 1dose, 0.2mL) 21days apart and administered IM.
  But, a third dose may be given at least 28 days after the second dose to individuals who are severely immunocompromised aged 5 to 11 years of age.
  Groups: Tozinameran (BNT162b2)
Biological: Tozinameran 6 months to 4 years of age — BNT162b2 (maroon cap) is administered with dilution by intramuscular injection (IM) of 0.2mL. According to the approved and authorized label, it is recommended that the recommended dose of BNT162b2 is administered by intramuscular injection (IM) twice (once a day, each 0.2mL) at least of 21 days apart, and Dose 3 at least 8 weeks later.
  Children who will turn from 4 years to 5 years of age between their doses in the vaccination course should receive their age-appropriate dose at the time of the vaccination and the interval between doses is determined by the child's age at the start of the vaccination course.
  The interchangeability of BNT162b2 with COVID-19 vaccines from other manufacturers to complete the vaccination course has not been established.
  BNT162b2 (6 months to 4 years of age) should be used only for infants and children 6 months to 4 years of age.
  Groups: Tozinameran (BNT162b2)
Biological: Riltozinameran 12 Years of age and older — The bivalent COVID-19 Vaccine for omicron (BA. 1) (grey cap) is administered by intramuscular injection (IM) of 0.3mL. There should be an interval of at least 3 months between administration of the bivalent COVID-19 Vaccine for omicron (BA. 1) and the last prior dose of a COVID-19 vaccine.
  The bivalent COVID-19 Vaccine for omicron (BA. 1) is only indicated for individuals who have previously received at least a primary vaccination course against COVID-19.
  Groups: Riltozinameran (BNT162b2 OMI BA.1)
Biological: Famtozinameran 12 Years of age and older — The bivalent COVID-19 Vaccine for omicron (BA. 4-5) (grey cap) is administered by intramuscular injection (IM) of 0.3mL. There should be an interval of at least 3 months between administration of the bivalent COVID-19 Vaccine for omicron (BA. 4-5) and the last prior dose of a COVID-19 vaccine.
  The bivalent COVID-19 Vaccine for omicron (BA. 4-5) is only indicated for individuals who have previously received at least a primary vaccination course against COVID-19.
  Groups: Famtozinameran (BNT162b2 OMI BA.4-5)
Biological: Famtozinameran 5 to 11 Years of age — The bivalent COVID-19 Vaccine for omicron (BA. 4-5) for 5 to 11 years of age (orange cap) is administered after dilution by intramuscular injection (IM) of 0.2mL. There should be an interval of at least 3 months between administration of the bivalent COVID-19 Vaccine for omicron (BA. 4-5) for 5 to 11 years of age and the last prior dose of a COVID-19 vaccine.
  The bivalent COVID-19 Vaccine for omicron (BA. 4-5) for 5 to 11 years of age is only indicated for individuals who have previously received at least a primary vaccination course against COVID-19.
  Groups: Famtozinameran (BNT162b2 OMI BA.4-5)
Biological: Raxtozinameran 12 years of age and older — BNT162b2 OMI XBB.1.5 (grey cap) is administered intramuscularly as a single dose of 0.3 mL for individuals 12 years of age and older regardless of prior COVID-19 vaccination status.
  For individuals who have previously been vaccinated with a COVID-19 vaccine, BNT162b2 OMI XBB.1.5 should be administered at least 3 months after the most recent dose of a COVID-19 vaccine.
  Groups: Raxtozinameran (BNT162b2 OMI XBB.1.5)
Biological: Raxtozinameran 6 months to 4 years of age — BNT162b2 OMI XBB.1.5 (maroon cap) is administered intramuscularly after dilution. For infants and children 6 months to 4 years of age without history of completion of a COVID-19, each 0.2 mL of dose is administered for a total of three vaccinations. The second dose is administered 3 weeks after the first dose followed by a third dose administered at least 8 weeks after the second dose. For infants and children 6 months to 4 years of age with history of completion of a COVID-19 primary course or prior SARS CoV-2 infection, a single dose of 0.2 mL is administered.
  Groups: Raxtozinameran (BNT162b2 OMI XBB.1.5)

SUMMARY:
This study will collect information on the safety of BNT162b2 products for subjects who have been administered in a routine clinical practice from 05Mar2021 to 04Mar2027 in Korea, and will be conducted in accordance with the New Drug Re-Examination Guideline of the Ministry of Food and Drug Safety (MFDS).

DETAILED DESCRIPTION:
This is an open-label, non-comparative, non-interventional, prospective, and multi-center study conducted in Korean health care centers by accredited physicians (investigator). The study population is Korean subjects who are scheduled for COVID-19 vaccination. BNT162b2 products will be administered according to the "Dosage and Administration" of the approved labeling. There is no visit or activity mandated by this study. The investigator will collect data from the subject's medical records and patient (subject) report outcome (PRO), and record the information on each subject's case report form (CRF).

Pfizer Pharmaceuticals Korea will conclude a post-marketing surveillance agreement with an investigator site before performing the study. Investigators at the institution that sign the agreement should prepare the CRFs from all the subjects who this vaccine was administered to after the start date of the study.

Each investigator will sequentially enroll all subjects to whom BNT162b2 products is prescribed for the first time according to the local product document and who agree to participate in this study by signing the data privacy statement used in place of the informed consent form until the total requested cases per center are collected for this study.

An electronic diary will be used in this study to collect adverse events that occur after injection. Follow-up exams will be carried out from after the first injection to before the second injection, and from after the second injection to 28 days after the second injection. Those who received booster doses will be followed up for the 28 days from the date of the booster dose. For the follow-up adverse event CRF, either an application using the mobile phones of subjects or entry on a paper questionnaire may be selected. The CRF will be filled out every day after the first and second injections. If an application is used, it is automatically sent as an eCRF. If a paper questionnaire is used, the questionnaire filled out after the first injection is collected at the time of the visit for the second injection, and the questionnaires filled out after the second injection and booster dose are collected 28 days after the second injection and 28 days after the booster dose respectively by mail.

To promote the collection of adverse events after injection, a reminder may be given by phone about entering the information and the collection of the CRF to subjects who gave consent beforehand. If it is difficult to record CRF due to the subject, the occurrence of adverse events can be confirmed by phone.

Safety is the primary interest of this study, which will be assessed based on adverse events (AEs) that occur during 28 days from the date of the first, second and booster doses of BNT162b2.

ELIGIBILITY:
1. Inclusion criteria

Subjects must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Korean subjects who are eligible for administration of BNT162b2 products (Including bivalent COVID-19 Vaccines for omicron) according to the locally approved and authorized label (indication, age criteria etc.)
2. Evidence of a personally signed and dated data privacy statement indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study - Data privacy statement signed by the subjects and parents or legal representative for subjects aged under 19

2. Exclusion criteria Subjects meeting any of the following criteria will be excluded in the study

1. Subjects who involved in the contraindications of use indicated in the locally approved and authorized label
2. Subjects with a history of hypersensitivity to any ingredients of this product or this product

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: the subjects who received the BNT162b2 under an approved label for use in Korea in contracted study sites.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2026-04-04 (Estimated); Study Completion 2026-04-04 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with Solicited adverse events | 1 week after administration of BNT162b2 products
  Solicited adverse events within 1 week (Day 1-7) after each dose of BNT162b2 products, and a number of subjects with such events will be collected.
Number of subjects with Unsolicited adverse events | 28 days after administration of BNT162b2 products
  Unsolicited adverse events within 28 days by its last dose, and a number of subjects with such events will be collected

SECONDARY OUTCOMES:
Number of subjects with Adverse Events (AEs) | 28 days after administration of BNT162b2 products
  All adverse events within 28 days by its last dose, and a number of subjects with such events will be collected
Number of subjects with Serious Adverse Events | 28 days after administration of BNT162b2 products
  All Serious adverse events within 28 days by its last dose, and a number of subjects with such events will be collected
Number of subjects with Expected Adverse Events | 28 days after administration of BNT162b2 products
  All expected adverse events within 28 days by its last dose, and a number of subjects with such events will be collected
Number of subjects with Adverse Drug Reactions | 28 days after administration of BNT162b2 products
  All adverse Drug Reactions within 28 days by its last dose, and a number of subjects with such events will be collected
Number of subjects with Serious Adverse Drug Reactions | 28 days after administration of BNT162b2 products
  All serious adverse drug reactions within 28 days by its last dose, and a number of subjects with such events will be collected
Number of subjects with Expected Adverse Drug Reactions | 28 days after administration of BNT162b2 products
  All expected adverse drug reactions within 28 days by its last dose, and a number of subjects with such events will be collected
Number of subjects with Unexpected Adverse Drug Reactions | 28 days after administration of BNT162b2 products
  All unexpected adverse drug reactions within 28 days by its last dose, and a number of subjects with such events will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591025